CLINICAL TRIAL: NCT01979081
Title: Detecting and Addressing Preclinical Disability
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Other Study IDs: Labarge 2013-02
Record Dates: First submitted 2013-05-14; First posted 2013-11-08 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Back Pain; Coronary Artery Disease; Chronic Obstructive Pulmonary Disease; Diabetes; Hypertension; Multiple Sclerosis; Osteoporosis; Osteoarthritis; Rheumatoid Arthritis; Stroke
MeSH Terms: conditions — Back Pain; Coronary Artery Disease; Pulmonary Disease, Chronic Obstructive; Diabetes Mellitus; Hypertension; Multiple Sclerosis; Osteoporosis; Osteoarthritis; Arthritis, Rheumatoid; Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- People with chronic disease: Participants greater than or equal to 44 years of age with a chronic disease (diabetes, heart disease, stroke, hypertension, osteoporosis, osteoarthritis, rheumatoid arthritis, chronic obstructive pulmonary disease, back pain, Multiple Sclerosis, Parkinson's Disease).
  Interventions: Other: Tailored advice from a physiotherapist and/or an occupational therapist through the myOSCAR patient portal
- People without chronic disease: Participants greater than or equal to 65 years of age without a chronic disease.
  Interventions: Other: Tailored advice from a physiotherapist and/or an occupational therapist through the myOSCAR patient portal

INTERVENTIONS:
Other: Tailored advice from a physiotherapist and/or an occupational therapist through the myOSCAR patient portal

SUMMARY:
The Physical Functioning Inventory (PFI) is a standardized patient reported outcome measure that assesses preclinical disability. Preclinical disability is a functional state in which people are still able to complete daily living tasks (e.g., walking, bathing) but are changing the frequency or modifying the way that they complete the tasks. The investigators have done some preliminary research using the PFI as an online monitoring tool (Richardson 2012), but further study is required to examine its psychometric properties and its suitability for use as a primary outcome measure. This measurement study has been designed to identify the optimal number of items on the PFI and to determine the reliability, validity, and responsiveness of the PFI when administered to a sample of adults and older adults both with and without chronic conditions. This project will also allow us to evaluate the use of self-monitoring of physical function and the added value of rehabilitation professionals to support self-monitoring. Using the results of the PFI, the investigators aim to develop a "tailored" population-based rehabilitation self-management intervention delivered through a secure messaging system in the patient's electronic personal health record (myOSCAR) that focuses on the early detection and prevention of preclinical disability.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 44 years of age
* Able to communicate in English
* Have had at least 3 physician visits in the last year
* Are able to access an email address independently
* Have a chronic disease

Exclusion Criteria:

* Any evidence of cognitive impairment
* Unable to travel to the clinic
* Awaiting long-term care
* Planning to relocate
* Experiencing an acute illness
* Are receiving palliative care

Ages: 44 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care center
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2013-01; Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Physical Functioning Inventory | Baseline, 3-5 days later, 6 months, 12 months, 18 months, 3-5 days later
  The PFI will be administered at baseline, then again 3-5 days later to assess test-retest reliability. It will then be administered at 6 months, 12 months and 18 months to determine its longitudinal validity. It will be administered a final time 3-5 days after the 18 month time frame to re-evaluate the measures test-retest reliability.

SECONDARY OUTCOMES:
Mobility Survey | Baseline, 3-5 days later, 6 months, 12 months, 18 months, 3-5 days later
  The Mobility Survey has been created from work by Manty (2007). Self-reported mobility is determined by asking participants to rate their ability to walk 2.0km, walk 0.5km, and climb up 1 flight of stairs on a scale of 1 (able to manage without difficulty) to 5 (unable to manage even with help). To identify persons at an early stage of mobility limitation (preclinical mobility limitation), additional questions were posed to participants who reported no task difficulty. The questions concerned the modification of task performance and the alternatives given were resting in the middle of the performance, using an aid, taking support from handrails, having reduced the frequency of performing the task, having slowed down performance of the task, experiencing tiredness when performing the task, or some other change in carrying out the task.
The Rapid Assessment of Physical Activity (RAPA) | Baseline, 3-5 days later, 6 months, 12 months, 18 months, 3-5 days later
Patient Specific Functional Scale (PSFS) | Baseline, 18 months
  The participant is asked to identify up to 5 important activities that they are unable to do or have difficulty with because of their health. For each of the activities the participant is asked to rate their ability to perform that activity on a scale of 0 (unable to perform the activity) to 10 (able to perform the activity like I always have).

OTHER OUTCOMES:
Center for Epidemiological Studies Depression Scale (CESD-R) | Baseline, 18 months
Brief Pain Inventory | Baseline, 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Julie Richardson, PhD, Principal Investigator — McMaster University; Lori Letts, PhD, Principal Investigator — McMaster University
Locations (1):
- Stonechurch Family Health Centre, Hamilton, Ontario, Canada